CLINICAL TRIAL: NCT04884074
Title: Effect of Routine Anterior Crural Repair in De-Novo Gastroesophageal Reflux After Laparoscopic Sleeve Gastrectomy - A Randomized Control Trial
Brief Title: Effect of Routine Anterior Crural Repair in De-Novo Gastroesophageal Reflux After Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Enders K.W. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRE-2016.202
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Gastro Esophageal Reflux Disease
Keywords: Obesity; Gastro Esophageal Reflux Disease; Laparoscopic Sleeve Gastrectomy; Anterior Crural Repair
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Intervention Model Description: Randomized double-blind controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization is done by telephone call to the randomization centre where a dedicated research assistant without detailed knowledge of the recruited patient's background will open a sealed envelope containing a computer-generated random number which indicates the mode of intervention. Both the patients and clinical assessors (independent of the operating surgeons) are blind to the mode of intervention in the first one year of enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): The procedure done to this group is Sleeve Gastrectomy with Anterior Crural Repair (ACR)
  Interventions: Procedure: Standard Sleeve Gastrectomy plus Anterior Crural Repair
- The control group (Other): The procedure done to this group is the Standard Sleeve Gastrectomy (SSG)
  Interventions: Procedure: Standard sleeve gastrectomy (SSG, the control group)

INTERVENTIONS:
Procedure: Standard Sleeve Gastrectomy plus Anterior Crural Repair — The procedure is performed in a similar fashion as standard sleeve gastrectomy. After gastric mobilization is completed as standard sleeve gastrectomy, the anterior phrenoesophageal ligament is divided and distal 3cm esophagus is mobilized. A Mid-Sleeve tube (40Fr) is inserted per-orally by the anesthetist and the hiatus opening is closed with 2/0 non-absorbable suture over the bougie anterior to the esophagus. The hiatus repair was sized by comfortably placement a dissection forceps adjacent to the esophagus without tension. Sleeve gastrectomy is then performed as the standard technique.
  Arms: The study group
Procedure: Standard sleeve gastrectomy (SSG, the control group) — The procedure is performed in French position with a standard 5-port approach and a pneumoperitoneum not exceeding 15mmHg.
  The greater omentum is then completely detached from the greater curvature of stomach using either ultrasonic or bipolar shear device. All adhesion between posterior gastric wall and pancreatic capsule is freed and the cardia is completely free with left crura completely exposed. A Mid-Sleeve tube (40Fr) is inserted per-orally by the anesthetist with its balloon tip reaching the gastric antrum and insufflated with 50cc of air. Sleeve gastrectomy is then performed using laparoscopic linear staplers, starting from a point 5-6cm proximal to the pylorus up cardia at about 1cm lateral to the angle of His, along the Mid-sleeve tube which is lying against the lesser curve of stomach. The staple line is reinforced with absorbable sutures. Distal stomach is anchored at retroperitoneum with non-absorbable stitch.
  Arms: The control group

SUMMARY:
The purpose of the study is to evaluate the superiority of anterior crural repair during sleeve gastrectomy over no repair in decreasing the incidence of gastroesophageal reflux disease.

DETAILED DESCRIPTION:
Introduction Obesity is a global pandemic. The prevalence of overweight and obesity is increasing globally. Together with its co-morbidities, obesity substantially decreased quality of life and life expectancy. Bariatric surgery has been shown to provide substantial and sustained effects on weight loss and ameliorates obesity-related comorbidities. Among different bariatric procedures, laparoscopic sleeve gastrectomy (LSG) is increasingly being performed due to the favorable bariatric outcome, simplicity of the procedure and relatively low complication profile as compared to bypass procedure.

Development of gastroesophageal reflux disease (GERD is a major health concern after LSG. It has been observed in the bariatric surgical community that many patients are complaining of persisted GERD symptoms after LSG surgery.

Aiming to avoid post-operative GERD, hiatal dissection with crural repair had been suggested to be performed on top of the sleeve gastrectomy procedure.

Data Collection Baseline data collection: All potential candidates will be screened for secondary causes of obesity, such as hypothyroidism and Cushing's syndrome, and are assessed for severity of obesity-related diseases including hypertension, diabetes mellitus, obstructive sleep apnoea syndrome and hyperlipidaemia. Extensive counseling will be given and potential benefits and complications of treatments will be discussed with all participants at least 4 weeks prior to recruitment.

Procedure data: Operative time, blood loss and total hospital stay are captured prospectively. All peri-operative complications will be documented and graded according to the Clavien-Dindo Classification System to facilitate comparison.

Follow-up and assessment:

Patients will be followed up at a designated Multi-disciplinary Clinic of Metabolic and Bariatric Surgery at 4 weeks, 3 months, 6 months, 9 months and 1 year after the operation. A standard dietary and exercise regimen will be prescribed to the patients, and their compliance to the life-style modification is monitored by designated dietitians. Counselling will be provided whenever necessary.

They are assessed for symptomatology according to a standard checklist by independent assessors who are blind to the mode of surgery performed. Data collection and blood tests, endoscopy and esophageal function test (see below) will be carried out during clinic visits.

Adherence to Good Clinical Practices (GCPs) This trial will reference the international ethical principles endorsed by the World Medical Association Declaration of Helsinki as well as ICH/GCP Standards, and any other applicable local laws or regulations

Data Completion and Record Keeping The hard-copy of patients' medical records will be kept in the Prince of Wales Hospital and the electronic information regarding patient information will be stored in the University/Hospital computer and password encrypted. Only the principle investigator, co-investigator and the research nurse will have the right to access these data. Data will be stored for 5 years and after completion of study, both hard & soft copy of the patients & study data will be destroyed and deleted of a body function or damage to a body structure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject without previous bariatric procedure and meets IFSO Asia-Pacific Chapter Consensus of Metabolic & Bariatric surgery criteria:

   i. BMI more than 35 kg/m2 with or without co-morbidities. ii. BMI more than 30 kg/m2 with obesity related co-morbidities.
2. Subject without evidence of gastroesophageal reflux disease i. Symptomatic - No gastroesophageal reflux symptom (GerdQ score no greater than 7) ii. Endoscopic - No esophagitis. No Hiatus Hernia (apparent separation distance between the squamocolumnar junction and the diaphragmatic impression greater than 2 cm) iii. Functional

1. High-resolution manometry 2. 24-hour esophageal pH study 4. ASA Class I - III 5. Subject is willing to give consent and comply with evaluation and treatment scheduled

Exclusion Criteria:

1. Pre-existing GERD, evident symptomatically, endoscopically or upon functional testing
2. Presence of Hiatus hernia (>2cm) or esophagitis
3. Previous upper GI surgery (e.g. bariatric surgery, anti-reflux surgery; gastrectomy; esophageal surgery)
4. Underlying uncontrolled endocrine problem that lead to obesity. (e.g. Hypothyroidism, Cushing syndrome, eating disorder etc)
5. ASA grade IV & V
6. Mental or psychiatric disorder; Drug or alcohol addiction
7. Cirrhosis or portal hypertension
8. Pregnant or breast feeding
9. Any condition which precludes compliance with the study;
10. History or presence of pre-existing autoimmune connective tissue disease
11. Active malignant disease. Patients with malignant disease who have been disease-free for at least 5 years are eligible
12. Active infection
13. Life expectancy less than 12 months
14. Special population, e.g. prisoner, mentally disabled, investigators' student or employees

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic GERD | 1 year
  Defined by GerdQ score > 7

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Suter M, Dorta G, Giusti V, Calmes JM. Gastro-esophageal reflux and esophageal motility disorders in morbidly obese patients. Obes Surg. 2004 Aug;14(7):959-66. doi: 10.1381/0960892041719581. PMID 15329186
- [Background] Mahawar KK, Jennings N, Balupuri S, Small PK. Sleeve gastrectomy and gastro-oesophageal reflux disease: a complex relationship. Obes Surg. 2013 Jul;23(7):987-91. doi: 10.1007/s11695-013-0899-x. PMID 23460263
- [Background] Tai CM, Huang CK. Increase in gastroesophageal reflux disease symptoms and erosive esophagitis 1 year after laparoscopic sleeve gastrectomy among obese adults. Surg Endosc. 2013 Oct;27(10):3937. doi: 10.1007/s00464-013-3022-4. Epub 2013 May 25. No abstract available. PMID 23708727
- [Background] Daes J, Jimenez ME, Said N, Dennis R. Improvement of gastroesophageal reflux symptoms after standardized laparoscopic sleeve gastrectomy. Obes Surg. 2014 Apr;24(4):536-40. doi: 10.1007/s11695-013-1117-6. PMID 24203681
- [Background] Wong SK, Lok H, Lam CC, Ng EK. Small Hiatus Hernia and Gastroesophgeal Reflux after Laparoscopic Sleeve Gastrectomy in Morbidly Obese Chinese. Obes Surg. 2014;24(8):1243.